CLINICAL TRIAL: NCT00260611
Title: Study of Oxaliplatin and Taxotere in Androgen Independent Prostate Cancer
Brief Title: Study of Oxaliplatin and Taxotere in Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 04-011
Record Dates: First submitted 2005-11-29; First posted 2005-12-01 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2015-03

CONDITIONS: Prostate Cancer
Keywords: prostate
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Oxaliplatin; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Oxaliplatin and Taxotere (Experimental): Patients will receive both docetaxel and oxaliplatin, IV on day 1 of each cycle. Treatment will be repeated every 21 days for up to 6 courses in the absence of disease progression, unacceptable toxicity, or >50% increase in serum PSA.
  Interventions: Drug: Oxaliplatin; Drug: Taxotere

INTERVENTIONS:
Drug: Oxaliplatin
  Other Names: eloxatin
Drug: Taxotere
  Other Names: Docefrez; Docetaxel

SUMMARY:
The primary objective for this study is to evaluate PSA response rates (response will be defined as a > 50% reduction in PSA levels) in men who have failed primary chemotherapy. The secondary objectives are to compare progression free survival, disease free survival, overall survival, and toxicity (tolerance/safety).

DETAILED DESCRIPTION:
This is a single institution phase II study of oxaliplatin and Taxotere in patients with androgen independent prostate cancer previously treated with up to two cytotoxic chemotherapy regimens. During this study, the efficacy and safety of this combination will be evaluated. The primary objective for this study is to evaluate PSA response rates (response will be defined as a > 50% reduction in PSA levels) in men who have failed primary chemotherapy. The secondary objectives are to compare progression free survival, disease free survival, overall survival, and toxicity (tolerance/safety). There will be up to 35 male subjects >= 18 years of age enrolled on this single institution study.

ELIGIBILITY:
Inclusion Criteria:

Must have histologically or cytologically confirmed adenocarcinoma consistent clinically and histologically with carcinoma of the prostate Confirmed androgen independent prostate cancer (progression despite castrate levels of serum testosterone) Measurable or evaluable disease (PSA elevation will constitute evaluable disease) 18 years of age. Because no dosing or adverse event data are currently available on the use of oxaliplatin in patients < 18 years of age, they are excluded from this study.

Life expectancy of greater than 3 months. ECOG Performance status of 0-1. No more than 2 prior regimens of cytotoxic chemotherapy. Androgen deprivation (castration or LHRH analogue), and prior antiandrogens allowed.

Patients must be off bicalutamide or nilutamide > 42 days, megestrol or flutamide > 28 days.

Concurrent bisphosphonate therapy allowed. Patients with prior radiotherapy for treatment of their bony metastases will be included if time since radiation is > 4 weeks, and if PSA is clearly rising.

Patients must have acceptable organ function as defined as: :WBC > 2500/mm3 or ANC > 1500/mm3, hemoglobin > 9.0 g/dL, platelet count > 100,000/mm3; Bilirubin < 1.5 mg/dL, SGOT/SGPT < 2 x ULN (< 4 x ULN if liver metastases present), PT/PTT normal; Creatinine < 1.8 mg/dL Adequate neurologic function defined as no clinically significant peripheral neuropathy, defined as any neuropathy ≤ grade 1.

Adequate cardiovascular function defined as no active congestive heart failure, no uncontrolled angina, no myocardial infarction within the past 6 months.

Exclusion Criteria:

No other experimental treatment, cytotoxics or radiation 4 weeks prior to enrollment. May not be taking other investigational drugs while on trial.

Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.

No prior therapy with oxaliplatin is allowed. No history of allergic reactions attributed to the drugs used in this study or compounds of similar chemical or biologic composition.

No history of intolerance or allergy to the antiemetics to be administered in conjunction with the study drugs (i.e., 5 HT3 antagonists).

No concurrent other active cancer from another primary site, except squamous cell and basal cell carcinoma of the skin.

No other serious concomitant illness will be allowed, including interstitial pneumonia, extensive and symptomatic fibrosis of the lung, uncontrolled hypertension, unstable angina, symptomatic congestive heart failure, NYHA Class III or IV, serious cardiac arrhythmia, uncontrolled diabetes mellitus or active infection.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2004-11; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
To evaluate PSA response rates (response will be defined as a > 50% reduction in PSA levels) in men who have failed primary chemotherapy. | Followed for survival
  Subjects once off treatment wil be followed for survival

SECONDARY OUTCOMES:
To compare progression free survival, disease free survival, overall survival, and toxicity (tolerance/safety). | Follow for survival
  Subjects will be followed for survival

CONTACTS AND LOCATIONS:
Overall Officials: Leonard J Appleman, MD, Principal Investigator — University of Pittsburgh Medical Center
Locations (1):
- Hillman Cancer Center, Pittsburgh, Pennsylvania, United States